CLINICAL TRIAL: NCT02274051
Title: The Safety and Tolerability of Kinetin, a Nutritional Supplement That Corrects the Splicing Defect, in Patients With Familial Dysautonomia
Brief Title: The Safety and Tolerability of Kinetin, in Patients With Familial Dysautonomia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0762
Record Dates: First submitted 2014-10-21; First posted 2014-10-24 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Familial Dysautonomia
MeSH Terms: conditions — Dysautonomia, Familial | interventions — Kinetin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kinetin (Experimental): Kinetin titration phase to 30mg/kg dose or individual max dose taken once daily.
  Patients will then proceed to steady state long-term phase at maximum individual dose of kinetin over a 3 year period.
  Interventions: Dietary Supplement: Kinetin

INTERVENTIONS:
Dietary Supplement: Kinetin — Titration of Kinetin to maximum individualized dose, then steady state over a 3 year period once daily dose.

SUMMARY:
This is a study of kinetin, a nutritional supplement that corrects the mRNA splicing defect in patients with familial dysautonomia (FD, also known as Riley Day syndrome or hereditary sensory and autonomic neuropathy type III). FD is a rare fatal autosomal recessive disease in which the growth and development of selective neuronal populations is impaired. The disease is the result of a point mutation in the gene sequence that encodes for kinase complex associated protein (IKAP) in chromosome 9q31. The mutation, at the start of the non-encoding intron 20, weakens the splice site, causing the spliceosome to wrongly join together exons 19 and 21 when transcribing the mRNA strand and miss out exon 20. The mutated mRNA produces a short unstable IKAP protein that is quickly degraded. Interestingly, the mutation does not lead to a complete loss of function. Instead, it results in a tissue specific deficiency in splicing efficiency with both normal (wild type) and mutant IKAP mRNA being expressed in different ratios in different tissues. Some cells, like fibroblasts, produce mostly normal mRNA and protein, where as others, like neurons, produce mostly mutant mRNA and almost no functional protein product.

DETAILED DESCRIPTION:
Familial dysautonomia (FD, also called Riley Day syndrome or hereditary sensory and autonomic neuropathy type III) is an autosomal recessive disease caused by a point mutation in the kinase complex associated protein (IKAP) gene sequence (1, 2). This leads to a tissue specific splicing defect with variable "skipping" of exon 20 (1, 3, 4). The consequence is a devastating congenital sensory neuropathy, affecting pain and temperature perception (5) as well as afferent information from the viscera (6). As a result, patients suffer recurrent aspiration pneumonias, respiratory insufficiency, proprioceptive ataxia, scoliosis and the long-term consequences of volatile blood pressure including renal failure (7) and left ventricular hypertrophy (8).

In-vitro studies have shown that the plant hormone kinetin corrects the splicing defect and increases the production of normal IKAP protein levels in FD derived cell lines (9, 10). Preliminary studies in heterozygous carriers of the IKAP mutation showed that dietary supplementation with kinetin increased the production of correctly spliced IKAP mRNA, in white blood cells (11). Preliminary studies in patients with FD have demonstrated that kinetin also increases the expression of correctly spliced IKAP mRNA extracted from white blood cells. However, the effect of kinetin on mRNA levels in neuronal tissue is unknown.

The overall objective of this study is to assess the safety and tolerability of administering kinetin in patients with FD. The specific aim of this proposal is to determine the safety of a once daily dose of kinetin in patients with FD using a dose ascending titration and to determine the long-term safety and tolerability during 3-years of receiving a maximum tolerated steady state dose of kinetin. The investigators hope to also demonstrate early proof of concept that kinetin enhances the ability of neuronal tissue to correctly splice IKAP mRNA.

ELIGIBILITY:
Inclusion Criteria:

1. Male of female patients aged 16 and older
2. Confirmed diagnosis of familial dysautonomia by genetic testing
3. Written informed consent to participate in the trial and understanding that they can withdraw consent at anytime without affecting their future care.
4. Ability to comply with the requirements of the study procedures.

Exclusion Criteria:

1. Patients who have taken other nutritional supplements that may affect IKAP mRNA splicing within the last 30 days
2. Patients with a known hypersensitivity to any component of the nutritional supplement kinetin
3. Patients with atrial fibrillation, angina or an electrocardiogram documenting significant abnormality that may jeopardize the patient's health.
4. Patients with significant pulmonary, liver, renal (creatinine >2.5 mg/ml) or cardiac illness
5. Women who are pregnant or lactating
6. Women of childbearing potential who are not using medically accepted methods of contraception.
7. Patients who have a significant abnormality on clinical examination that may, in the investigator's opinion, jeopardize their healthy participating in this pilot trial.
8. Patients taking allopurinol, other xanthine oxidase inhibitors or other compounds that may interfere with the metabolism of kinetin including oral calcium supplements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-11; Primary Completion 2019-05-04 (Actual); Study Completion 2019-05-04 (Actual)

PRIMARY OUTCOMES:
Change in Safety blood labs | At baseline and after each 6 months period and at 36 months
  safety blood labs (CBC, metabolic panel)
Change in vital signs | At baseline and after each 6 months period and at 36 months
  Sitting and standing blood pressure measurements and heart rate
Change in ECG | At baseline and after each 6 months period and at 36 months
  12 lead ECG measures
Number of participants with adverse events | At baseline and after each 6 months period and at 36 months
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States